CLINICAL TRIAL: NCT07133217
Title: Comparative Evaluation of Postoperative Pain and Clinical Success Following Root Canal Treatment With Hand Files, ProTaper Ultimate, and WaveOne Gold Systems in Symptomatic Irreversible Pulpitis: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of Postoperative Pain and Clinical Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Kandemir Demirci, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-9.1/4; TS-GAP-2024-32255 (Other Grant/Funding Number: Ege University Scientific Research Projects)
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Bioceramic sealer; Clinical success; Emergency treatment; Hand file; Postoperative pain; Reciprocating file; Rotary file; Symptomatic irreversible pulpitis
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Preparation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Manuel Instrumentation Technique Group (Active Comparator): Root canals were prepared with hand files. Irrigation was performed with 10 mL of NaOCl, followed by 5 mL of 17% ethylenediaminetetraacetic acid (EDTA). Temporary coronal restoration was completed with glass ionomer cement. For this group, 72 hours after the completion of root canal preparation in the emergency intervention session, calcium hydroxide was applied to the root canals for 7 days, and the teeth were obturated using a bioceramic root canal sealer with the system-specific gutta-percha and obturation methods recommended by the manufacturers.
  Interventions: Device: Root canal preparation with Hand Files (Dentsply Sirona)
- Reciprocating Motion Technique Group (Active Comparator): Root canals were prepared with WaveOne Gold instruments and an X-Smart Plus (Dentsply Maillefer, Switzerland) endodontic motor. Irrigation was performed with 10 mL of NaOCl, followed by 5 mL of 17% ethylenediaminetetraacetic acid (EDTA). Temporary coronal restoration was completed with glass ionomer cement. For this group, 72 hours after the completion of root canal preparation in the emergency intervention session, calcium hydroxide was applied to the root canals for 7 days, and the teeth were obturated using a bioceramic root canal sealer with the system-specific gutta-percha and obturation methods recommended by the manufacturers.
  Interventions: Device: Root canal preparation with the WaveOne Gold file system (Dentsply Sirona, Ballaigues, Switzerland)
- Rotation Motion Technique Group (Active Comparator): Root canals were prepared with ProTaper Ultimate instruments and an X-Smart Plus (Dentsply Maillefer, Switzerland) endodontic motor. Irrigation was performed with 10 mL of NaOCl, followed by 5 mL of 17% ethylenediaminetetraacetic acid (EDTA). Temporary coronal restoration was completed with glass ionomer cement. For this group, 72 hours after the completion of root canal preparation in the emergency intervention session, calcium hydroxide was applied to the root canals for 7 days, and the teeth were obturated using a bioceramic root canal sealer with the system-specific gutta-percha and obturation methods recommended by the manufacturers.
  Interventions: Device: Root canal preparation with the ProTaper Ultimate file system (Dentsply Sirona)

INTERVENTIONS:
Device: Root canal preparation with Hand Files (Dentsply Sirona) — Root canal treatments were performed with hand files
  Arms: Conventional Manuel Instrumentation Technique Group
Device: Root canal preparation with the WaveOne Gold file system (Dentsply Sirona, Ballaigues, Switzerland) — Root canal treatments were performed with WaveOne Gold Files
  Arms: Reciprocating Motion Technique Group
Device: Root canal preparation with the ProTaper Ultimate file system (Dentsply Sirona) — Root canal treatments were performed with ProTaper Ultimate Files
  Arms: Rotation Motion Technique Group

SUMMARY:
Sixty-three mandibular molars with vital pulp, symptomatic acute pain, and a Numerical Rating Scale (NRS) score of 7 or higher-requiring emergency treatment-were randomly allocated into three groups according to the preparation systems to be used: conventional manual instrumentation technique with hand files, reciprocating motion technique with WaveOne Gold files, and rotary motion technique with ProTaper Ultimate files.

In the first session, patients received emergency treatment with one of the three file systems, and seven days later, root canal treatments were completed using the same system within each patient group. Preoperative pain scores of patients presenting to our clinic with acute pain were recorded using the Numerical Rating Scale (NRS).

During the emergency root canal treatment session, the first group was instrumented with hand files, the second group with WaveOne Gold files, and the third group with ProTaper Ultimate files, and the emergency treatment session was completed. Shaping times were measured during the procedures.

Following the emergency session, patients were instructed to record their postoperative pain at the 6th hour, 12th hour, and on the 1st, 2nd, 3rd, 4th, 5th, 6th, and 7th days using the provided NRS.

One week after the emergency treatment session, root canal obturation was performed using each system's own gutta-percha and Bioceramic root canal sealer. Clinical and radiographic follow-ups were carried out at 6 and 12 months.

DETAILED DESCRIPTION:
• This randomized clinical study was conducted to evaluate and compare the effects of the conventional step-back technique with hand files, the reciprocal technique with WaveOne Gold files, and the rotary technique with ProTaper Ultimate files on the frequency and intensity of pain before and after emergency treatment, as well as on clinical and radiological outcomes in symptomatic and acutely painful vital molars during root canal treatment.

Sixty-three symptomatic mandibular molars with vital pulp were randomly allocated into three groups according to the preparation system used: Hand files, WaveOne Gold, and ProTaper Ultimate. The file systems assigned to each group were used for root canal preparation in all cases.

In the rotary and reciprocating file groups, obturation was performed with their own gutta-percha using the single cone technique with Bioceramic sealer and in the conventional hand file group root canal obturation was performed with cold lateral compaction method.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* Patients who can come to regular check-ups and have high treatment motivation
* Patients who can establish an appropriate patient-doctor dialogue
* Patients without systemic disease
* Patients with teeth that have not previously undergone endodontic treatment
* Patients who meet the clinical definition of symptomatic irreversible pulpitis (pain, prolonged sensitivity to hot and cold,percussion sensitivity, pulpal bleeding)
* Delayed positive response of teeth to cold testing and electric pulp testing
* Presence of spontaneous pain before treatment
* Mandibular first or second molar with complete root development
* Formation of large pulpal perforation during caries removing
* Presence of bleeding in the exposed pulp that cannot be stopped within 5 minutes after the pulp exposure

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients at medical risk (patients with immune system diseases/systemic diseases, patients using medication),
* Patients with NSAID (non-steroidal anti-inflammatory) allergy
* Patients with allergy to the materials used during root canal treatment
* Patients who used antibiotics or analgesics before applying to the clinic
* Pregnant patients
* Asymptomatic or devital teeth
* Presence of advanced periodontal disease (probing depth> 3 mm)
* Patients with more than one tooth requiring endodontic treatment
* The relevant tooth has previously undergone endodontic treatment
* The tooth needs a post-core or is a prosthetic support tooth
* Presence of calcified root canal
* Teeth with internal or external root resorption
* Teeth with open apex
* Mandibular third molars

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
The incidence and intensity of post-obturation pain | up to 30-day
  Post-obturation pain up to 30 days after root canal treatment was measured with Numerical Rating Scale. The Numerical Rating Scale is a pain measurement scale that encompasses the following grades: 0 no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain.

SECONDARY OUTCOMES:
Clinical and radiographical success | Up to 1 year follow up
  Clinical success was determined by the absence of any clinical or radiographic indicators of inflammation or infection, and outcomes were categorized as either successful or unsuccessful.Unsuccessful ones were scored as "0" and successful ones as "1". During the clinical examination, the presence of swelling, pain, sinus tract formation, or tenderness upon percussion or palpation was documented. Periodontal probing depths were assessed for each case. Radiographic analysis evaluated the integrity of periodontal tissues and the presence or absence of periapical radiolucent areas. The level of root canal fillings was classified as short (≥2 mm from the apex), acceptable (0-2 mm), or overfilled (beyond apex).

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Kandemir Demirci, Associate Professor, Principal Investigator — Ege University Faculty of Dentistry
Locations (1):
- Gözde Kandemir Demirci, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No